CLINICAL TRIAL: NCT05510505
Title: A Prospective, Randomized, Multi-center Study to Assess the Efficacy and Safety of GVHD Prophylaxis by Addition of CD20 Monoclonal Antibody to the Conditioning Regimen in Severe Aplastic Anemia Patients With Treatment of Allogeneic HSCT
Brief Title: GVHD Prophylaxis by Addition of CD20 Monoclonal Antibody to the Conditioning Regimen in SAA With Treatment of Allo-HSCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Wu Depei, Professor, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAA-HSCT-2021
Record Dates: First submitted 2022-08-08; First posted 2022-08-22 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — 188Re-anti-CD20 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATG arm (control group) (Active Comparator): 4.2.1 Matched sibling donor 1) ATG arm (control group) Fludarabine 30mg/m2/d×6d（-7d ~ -2d）+ Cyclophosphamide 50mg/kg/d×2d （-4d ~ -3d）+ ATG 2.5mg/kg/d×5d（-8d ~ -4d）
  4.2.2 Unrelated donor and haploidentical donor
  1) ATG arm (control group) Busulfan 3.2 mg/kg/d（0.8 mg/kg，q6h）×2d（-7d ~ -6d） + Cyclophosphamide 50mg/kg/d×4d （-5d ~ -2d）+ ATG 2.5mg/kg/d×4d（-5d ~ -2d）
  Interventions: Drug: ATG
- ATG + CD20 monoclonal antibody (test arm) (Experimental): 4.2.1 Matched sibling donor 2) ATG + CD20 monoclonal antibody (test arm) Fludarabine 30mg/m2/d×6d（-7d ~ -2d） + Cyclophosphamide 50mg/kg/d×2d （-4d ~ -3d）+ ATG 2.5mg/kg/d×5d（-8d ~ -4d）+ CD20 monoclonal antibody 375mg/m2, -1d
  4.2.2 Unrelated donor and haploidentical donor 2) ATG + CD20 monoclonal antibody (test arm) Busulfan 3.2 mg/kg/d（0.8 mg/kg，q6h）×2d（-7d ~ -6d） + Cyclophosphamide 50mg/kg/d×4d （-5d ~ -2d）+ ATG 2.5mg/kg/d×4d（-5d ~ -2d）+ CD20 monoclonal antibody 375mg/m2, -1d
  Interventions: Drug: CD20 monoclonal antibody

INTERVENTIONS:
Drug: CD20 monoclonal antibody — 4.2 Conditioning Regimen
  4.2.1 Matched sibling donor
  1. ATG arm (control group) Fludarabine 30mg/m2/d×6d（-7d ~ -2d）+ Cyclophosphamide 50mg/kg/d×2d （-4d ~ -3d）+ ATG 2.5mg/kg/d×5d（-8d ~ -4d）
  2. ATG + CD20 monoclonal antibody (test arm) Fludarabine 30mg/m2/d×6d（-7d ~ -2d） + Cyclophosphamide 50mg/kg/d×2d （-4d ~ -3d）+ ATG 2.5mg/kg/d×5d（-8d ~ -4d）+ CD20 monoclonal antibody 375mg/m2, -1d
  4.2.2 Unrelated donor and haploidentical donor
  1. ATG arm (control group) Busulfan 3.2 mg/kg/d（0.8 mg/kg，q6h）×2d（-7d ~ -6d） + Cyclophosphamide 50mg/kg/d×4d （-5d ~ -2d）+ ATG 2.5mg/kg/d×4d（-5d ~ -2d）
  2. ATG + CD20 monoclonal antibody (test arm) Busulfan 3.2 mg/kg/d（0.8 mg/kg，q6h）×2d（-7d ~ -6d） + Cyclophosphamide 50mg/kg/d×4d （-5d ~ -2d）+ ATG 2.5mg/kg/d×4d（-5d ~ -2d）+ CD20 monoclonal antibody 375mg/m2, -1d
  Other Names: allogeneic hematopoietic stem cell transplantation
  Arms: ATG + CD20 monoclonal antibody (test arm)
Drug: ATG — 4.2 Conditioning Regimen
  4.2.1 Matched sibling donor
  1. ATG arm (control group) Fludarabine 30mg/m2/d×6d（-7d ~ -2d）+ Cyclophosphamide 50mg/kg/d×2d （-4d ~ -3d）+ ATG 2.5mg/kg/d×5d（-8d ~ -4d）
  2. ATG + CD20 monoclonal antibody (test arm) Fludarabine 30mg/m2/d×6d（-7d ~ -2d） + Cyclophosphamide 50mg/kg/d×2d （-4d ~ -3d）+ ATG 2.5mg/kg/d×5d（-8d ~ -4d）+ CD20 monoclonal antibody 375mg/m2, -1d
  4.2.2 Unrelated donor and haploidentical donor
  1. ATG arm (control group) Busulfan 3.2 mg/kg/d（0.8 mg/kg，q6h）×2d（-7d ~ -6d） + Cyclophosphamide 50mg/kg/d×4d （-5d ~ -2d）+ ATG 2.5mg/kg/d×4d（-5d ~ -2d）
  2. ATG + CD20 monoclonal antibody (test arm) Busulfan 3.2 mg/kg/d（0.8 mg/kg，q6h）×2d（-7d ~ -6d） + Cyclophosphamide 50mg/kg/d×4d （-5d ~ -2d）+ ATG 2.5mg/kg/d×4d（-5d ~ -2d）+ CD20 monoclonal antibody 375mg/m2, -1d
  Arms: ATG arm (control group)

SUMMARY:
Objectives 2.1 Primary objectives

1) To observe and compare incidence and severity of aGVHD and cGVHD between the two arms within 2 years after transplantation.

2) To observe and compare the engraftment rate between the two arms. 3) To observe and compare the incidence of infections between the two arms. 2.2 Secondary objectives

1. To conduct pharmacogenomic assay in CD20 arm(treatment arm) before conditioning and monitor plasma concentration of CD20 dynamically（7d、14d、28d、56d、91d）.
2. To monitor levels of B cells in peripheral blood dynamically (+90d、+180d、+270d、+360d、+450d、+540d、+630d、+720d) in all patients.
3. To observe and compare the incidence of PTLD between the two arms.
4. To observe and compare immunoglobulin levels after transplantation in all patients.
5. To evaluate transplant-related mortality.
6. To evaluate the effect on hematopoietic reconstruction.

DETAILED DESCRIPTION:
3. Study design 3.1 Principle of design: prospective, randomized, control, open label 3.2 Subjects: patients with SAA undergoing allogeneic HSCT 3.3 Grouping: In this study, central randomization was used for random enrolment (1:1). After signing the informed consent, patients were randomized into rituximab conditioning group (test group) or non- rituximab conditioning group (control group). Treatment was assigned on a randomized basis according to a 1:1 ratio. The test group and the control group each will include 100 cases.

3.4 Study schedule: This clinical research is to be completed from September 2020 to September 2023.

1. Subject enrollment 36months
2. Transplantation to the end of follow-up 24months
3. Data collection and report writing 3months In total 63months

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for inclusion in this study must meet all of the following criteria:

  1. SAA characterized Bone marrow cellularity< 25%, or 25-50% with <30% residual hematopoietic cells and pancytopenia, with at least two of the following parameters in peripheral blood Absolute neutrophil count < 0.5*10E9/L Platelet count < 20*10E9/L Absolute reticulocyte count < 20*10E9/L
  2. ALL patients will undergo allo-HSCT.
  3. Subjects aged <50 years old with KPS performance status ≥70 at the same time.
  4. Aspartate aminotransferase (AST) , alanine aminotransferase (ALT) and alkaline phosphatase≤2 times the upper limit of normal (ULN). Blood urea nitrogen and Creatinine ≤1.25 times ULN.
  5. Cardiac function of subjects must meet all of the following requirements: ECG examination do not reveal any acute myocardial infarction, arrhythmia, or first-degree or higher atrioventricular block. No signs of heart failure. No carrying of active rheumatoid heart disease. Chest radiograph or physical examination do not indicate an enlarged heart.
  6. ALL subjects show none contraindication for allogeneic hematopoietic stem cell transplantation.
  7. Patients enrolled in the rituximab group have no contraindications for the use of rituximab.
  8. Patients and their clients are willing to perform hematopoietic stem cell transplantation.
  9. Potential donor is accessible.
  10. Patients have no anti-HLA antibodies.

Exclusion Criteria:

1. Subject who is unable comprehend or is unwilling to sign an informed consent form or consent form due to severe physical or mental illness resulting in a survival of less than 2 years.
2. Presence of clinically active uncontrolled significant chronic infections (including bacterial, fungal or viral infection), such as dental caries, otitis media, sinusitis, etc., need to be carried out after effective control.
3. Past medical history of severe pulmonary dysfunction.
4. Past medical history of diabetes with a propensity for ketoacidosis.
5. Presence of severe coagulopathy, thrombophlebitis or pulmonary embolism.
6. Presence of decompensated liver insufficiency or active hepatitis.
7. Presence of history of severe autoimmune disease.
8. Past medical history of thyroid dysfunction with currently abnormal thyroid function.
9. Any concomitant malignancies that have not been disease-free for 5 years.
10. Past medical history of hypersensitivity to biological products (including antibiotics).
11. Pregnant or nursing woman.
12. Inherited bone marrow failure.

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
GVHD incidence | 2 years
  GVHD incidence, location and grade. Infection incidence and recurrence rate.

SECONDARY OUTCOMES:
Infection incidence | 2 years
  Cumulative incidence of infection post-transplant
GVHD-free survival rate | 2 years
  defined by the percentage of patients who are alive without evidence of moderate or severe chronic GVHD at 2 year
transplant related mortality | 2 years
  Defined as the number of days from the date of transplant to the date of death related to transplant
overall survival rate | 2 years
  OS is defined as the number of days from the date of transplant to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: depei wu, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No